CLINICAL TRIAL: NCT05792332
Title: Integrated Management of Atypical Parkinsonism: A Home-based Patient-Centered Healthcare Delivery Based on Telenursing. A Multicenter, Interventional Non-pharmacological, Randomized, Single-blind Clinical Trial. IMPACT Study
Brief Title: Integrated Management of Atypical Parkinsonism: A Home-based Patient-Centered Healthcare Delivery Based on Telenursing (IMPACT Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Fondazione Mondino (Other); Neuromed IRCCS (Other); Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IMPACT
Record Dates: First submitted 2023-02-24; First posted 2023-03-31 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Atypical Parkinsonism; MSA - Multiple System Atrophy; PSP; Nurse-Patient Relations; Nurse Physician Relations
Keywords: Atypical parkinsonism; Nurse Specialist; MSA; PSP
MeSH Terms: conditions — Shy-Drager Syndrome | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Experimental): Patients are followed up by a nurse-telemonitoring
  Interventions: Other: Telemonitoring
- Standard-of-care (Active Comparator): Patients are followed up only by the neurologist
  Interventions: Other: Standard-of-care

INTERVENTIONS:
Other: Telemonitoring — Patients are followed up by a nurse specialist in parkinsonism who interacts with the treating neurologist and a multidisciplinary team
  Arms: Telemonitoring
Other: Standard-of-care — Patients are managed only by the neurologist according the institution's clinical practice
  Arms: Standard-of-care

SUMMARY:
This project aims to investigate whether an integrated model based on proactive and reactive telenursing monitoring coordinated by a parkinsonism nurse specialist (case manager) is able to improve care delivery and quality of life of patients with atypical parkinsonisms. This could reduce the risk (e.g. through health education counselling) and the severity of complications (e.g. falls). Main responsibilities of the Co-PI: project idea and supervision, coordination of the study, patient selection and recruitment, patient recruitment, participation in statistical analysis and drafting the manuscript. Co-PI is responsible of the rate of recruitment and drop-out

DETAILED DESCRIPTION:
People with parkinsonism experience a wide range of motor and non-motor disorders associated with the increasing complexity of care delivery and the increased risk of complications with increased hospital access. Although a number of multidisciplinary care models have been proposed so far, results have been disappointing in terms of benefit in quality of life and cost-effectiveness. An integrated remote care model at home, involving a parkinsonism nurse specialist (PKNS) as well as a movement disorder specialist, could offer significant benefits to patients and healthcare professionals through better health education, continuity of care and more careful monitoring of the complications of the accident. In this multicenter, randomized, single-blinded, case-control trial, the investigators will recruit 164 patients with atypical parkinsonism (either MSA or PSP) to investigate the efficacy and cost-effectiveness of a 12-month remote home-based integrated program to improve healthcare delivery, coordinated by a specialized nurse (case manager) compared to standard medical care. This organizational model of personalized medicine aims to simplify, standardize and improve patient care and monitoring over time, including remote management of situations of urgency. This telenursing program consists of both proactive and reactive monitoring approaches acting synergistically to optimize the continuity of care by tertiary expert movement disorders clinics. In proactive monitoring, patients are contacted at baseline (to create a patient record focused on identifying individual-specific vulnerabilities) and then every 3 months. During the 12-month study period, patients and caregivers may contact the case manager in case of any problems (reactive monitoring), who may: (a) deal with the specific problem also by interacting with the participant's general practitioner and other healthcare professionals (e.g. physical therapist, psychologist, nutritionist, occupational therapist, social worker, etc) or (b) refer to the neurologist for teleconsultation or in-person visit according to a semi-structured algorithm, which assigns 4 levels of priority. Participants will be evaluated with clinical scales testing the quality of life, motor and non-motor symptoms, caregiver burden, adherence to therapy, cumulative disease burden and the number of unscheduled hospital access during the study period. The cost-effectiveness of this method will also be evaluated by using the EuroQoL, which will estimate the incremental cost per quality-adjusted life-years (QALY) gain. Finally, the investigators will assess the feasibility and utility of Telemonitoring to guide decisionmaking by using a waist-worn wearable (STAT-ONTM) to monitor real-life motor autonomy and the risk of falls, including freezing of gait for 5 consecutive days every month during the 12-month duration of the study. If successful, this low-cost integrated management of patients with atypical parkinsonism may be extended to people with the more prevalent Parkinson's disease as well as other neurodegenerative disorders (e.g. Alzheimer's dementia)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MSA or PSP in all their possible variants (MSA-P, MSA-C; PSP-RS, PSP-P, PSP-CBS, etc.) according to internationally validated criteria.

Exclusion Criteria:

* Hoehn and Yahr stage = 5 in ON phase
* Clinical Frialty Scale (CFS) ≥ 8
* Serious medical disorders that, in the opinion of the recruiting neurologist, may impair participation in the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Changes in total score of the Parkinson's Disease Questionnaire 39-items scale (PDQ-39) | baseline, week 52
  Thi is a 39-items questionnaire assessing the quality of life of patient with Parkinsonism. Score is expressed in percentage from 0% to 100%. The higher the score the lower the quality of life

SECONDARY OUTCOMES:
Changes in the Movement Disorder Society Unified Parkinson's Disease Rating Scale part II (MDS-UPDRS Part II) | baseline, week 52
  This is a scale (MDS-UPDRS Part II) used to assess activities of daily living. Score ranges from 0 to 52. The higher the score the worse the Disability
Changes in the Movement Disorder Society Unified Parkinson's Disease Rating Scale part IV (MDS-UPDRS part IV) | baseline, week 52
  This is a scale (MDS-UPDRS part IV) used to assess complications of dopaminergic therapy. Score ranges from 0 to 24. The higher the score the worse the disability
Changes in the Non-Motor Symptoms Scale score (NMSS) | baseline, week 52
  This is a scale used to assess the burden of non-motor symptoms in Parkinson's disease. Total score is 0-360. The higher the score the worse the disability
Changes in Unified Multiple System Atrophy Rating Scale (UMSARS) | baseline, week 52
  This scale (UMSARS) is used to assess disease progression in multiple system atrophy.The score is from 0 up to 109. The higher the score the worse the disability
Changes in Progressive Supranuclear Palsy Rating Scale (PSPRS) | baseline, week 52
  This scale (PSPRS) is used to assess disease progression in Progressive Supranuclear Palsy. The total score is 0-100. The higher the score the worse the disability
Changes in the activities of daily living questionnaire (ADL_questionnaire) | baseline, week 52
  The "ADL (Activities of Daily Living)" evaluation refers to the fundamental activities of daily life in which the subject is dependent: on a scale from 0 to 6 points, the lower the score, the greater the person's need for assistance
Changes in the intrumental activities of daily living questionnaire (IADL) | baseline, week 52
  The "IADL (Instrumental Activities of Daily Living)" evaluation refers to the instrumental activities of daily life in which the subject is dependent (eg using telephone, preparing meals, taking medications, etc): on a scale from 0 to 8 points, the lower the score, the greater the person's need for assistance
Changes in the Zarit Burden Interview scale score (ZBI) | baseline, week 52
  This is a scale used to investigate caregiver's burnout. Total score is 0-40. The higher the score the worse the disability
Number of unplanned hospital admission | week 52
  Sum of number of outpatients departments assessments, number of emergency rooms accesses, number of unplanned hospitalizations
Number of incident comorbidities | baseline, week 52
  The number of incident comorbidities over the 12.month study period will be assessed using a semistructured interview
Changes in Euro Quality Of Life Dimensions-5 Levels score (EuroQOL-5) | baseline, week 52
  This is a useful and validated instrument to measure quality of life in patients with Parkinson's disease. The patient select a score from 0 to 100. The lowest the score the lowest quality of life.
Changes in the Morisky Medical Adherence scale-8 items score (MMAS) | baseline, week 26, week 52
  This is an 8-items scale used to investigate patient adherence to the therapy prescribed by the MD specialist. Score is 0-8 "yes" answer. The 3 categorical Likert Scale is: low adherence <6; medium adherence 6-8; high adherence 8.
Changes in patient experience questionnaire (EQ) | baseline, week 26, week 52
  This is a questionnaire assessing patient perception and satisfaction of the quality of health care. Total score is 0-100. The highest the score, the worst the satisfaction
Changes in freezing of walking, Freezing of gait-questionnaire (FOG-Q) | baseline, week 52
  Changes in gait performances, mainly in freezing of walking, are analysis by this questionnaire. Total score is 0-24. The highest the score, the highest the freezing

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Eleopra, MD, Principal Investigator — Study Principal Investigator Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Universitaria Gaetano Martino, Messina
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Fondazione IRCCS Istituto Neurologico Nazionale Casmiro Mondino, Pavia
  - IRCCS Neuromed, Pozzilli

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest on this topic. Data shared will be coded, with no protected health information included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months.
  Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement. For more information or to submit a request, please contact crc@istituto-besta.it

REFERENCES:
- [Background] van der Marck MA, Bloem BR, Borm GF, Overeem S, Munneke M, Guttman M. Effectiveness of multidisciplinary care for Parkinson's disease: a randomized, controlled trial. Mov Disord. 2013 May;28(5):605-11. doi: 10.1002/mds.25194. Epub 2012 Nov 19. PMID 23165981
- [Background] Huse DM, Schulman K, Orsini L, Castelli-Haley J, Kennedy S, Lenhart G. Burden of illness in Parkinson's disease. Mov Disord. 2005 Nov;20(11):1449-54. doi: 10.1002/mds.20609. PMID 16007641
- [Background] Gerlach OH, Broen MP, van Domburg PH, Vermeij AJ, Weber WE. Deterioration of Parkinson's disease during hospitalization: survey of 684 patients. BMC Neurol. 2012 Mar 8;12:13. doi: 10.1186/1471-2377-12-13. PMID 22400982
- [Background] Muzerengi S, Herd C, Rick C, Clarke CE. A systematic review of interventions to reduce hospitalisation in Parkinson's disease. Parkinsonism Relat Disord. 2016 Mar;24:3-7. doi: 10.1016/j.parkreldis.2016.01.011. Epub 2016 Jan 13. PMID 26803377
- [Background] Hassan A, Wu SS, Schmidt P, Dai Y, Simuni T, Giladi N, Bloem BR, Malaty IA, Okun MS; NPF-QII Investigators. High rates and the risk factors for emergency room visits and hospitalization in Parkinson's disease. Parkinsonism Relat Disord. 2013 Nov;19(11):949-54. doi: 10.1016/j.parkreldis.2013.06.006. Epub 2013 Jul 5. PMID 23835430
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479
- [Background] Hagell P, Alvariza A, Westergren A, Arestedt K. Assessment of Burden Among Family Caregivers of People With Parkinson's Disease Using the Zarit Burden Interview. J Pain Symptom Manage. 2017 Feb;53(2):272-278. doi: 10.1016/j.jpainsymman.2016.09.007. Epub 2016 Nov 1. PMID 27810571
- [Background] Miller MD, Paradis CF, Houck PR, Mazumdar S, Stack JA, Rifai AH, Mulsant B, Reynolds CF 3rd. Rating chronic medical illness burden in geropsychiatric practice and research: application of the Cumulative Illness Rating Scale. Psychiatry Res. 1992 Mar;41(3):237-48. doi: 10.1016/0165-1781(92)90005-n. PMID 1594710
- [Background] Schrag A, Selai C, Jahanshahi M, Quinn NP. The EQ-5D--a generic quality of life measure-is a useful instrument to measure quality of life in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2000 Jul;69(1):67-73. doi: 10.1136/jnnp.69.1.67. PMID 10864606
- [Background] Fabbrini G, Abbruzzese G, Barone P, Antonini A, Tinazzi M, Castegnaro G, Rizzoli S, Morisky DE, Lessi P, Ceravolo R; REASON study group. Adherence to anti-Parkinson drug therapy in the "REASON" sample of Italian patients with Parkinson's disease: the linguistic validation of the Italian version of the "Morisky Medical Adherence Scale-8 items". Neurol Sci. 2013 Nov;34(11):2015-22. doi: 10.1007/s10072-013-1438-1. Epub 2013 Jun 1. PMID 23728715
- [Background] Wenning GK, Stankovic I, Vignatelli L, Fanciulli A, Calandra-Buonaura G, Seppi K, Palma JA, Meissner WG, Krismer F, Berg D, Cortelli P, Freeman R, Halliday G, Hoglinger G, Lang A, Ling H, Litvan I, Low P, Miki Y, Panicker J, Pellecchia MT, Quinn N, Sakakibara R, Stamelou M, Tolosa E, Tsuji S, Warner T, Poewe W, Kaufmann H. The Movement Disorder Society Criteria for the Diagnosis of Multiple System Atrophy. Mov Disord. 2022 Jun;37(6):1131-1148. doi: 10.1002/mds.29005. Epub 2022 Apr 21. PMID 35445419
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Borzi L, Mazzetta I, Zampogna A, Suppa A, Irrera F, Olmo G. Predicting Axial Impairment in Parkinson's Disease through a Single Inertial Sensor. Sensors (Basel). 2022 Jan 6;22(2):412. doi: 10.3390/s22020412. PMID 35062375
- [Background] Cilia R, Mancini F, Bloem BR, Eleopra R. Telemedicine for parkinsonism: A two-step model based on the COVID-19 experience in Milan, Italy. Parkinsonism Relat Disord. 2020 Jun;75:130-132. doi: 10.1016/j.parkreldis.2020.05.038. Epub 2020 Jun 10. PMID 32723588
- [Result] Lennaerts H, Groot M, Rood B, Gilissen K, Tulp H, van Wensen E, Munneke M, van Laar T, Bloem BR. A Guideline for Parkinson's Disease Nurse Specialists, with Recommendations for Clinical Practice. J Parkinsons Dis. 2017;7(4):749-754. doi: 10.3233/JPD-171195. PMID 28800338
- [Derived] Cilia R, Colucci F, Suppa A, Valentino F, Terranova C, Leuzzi C, Cordasco J, Fusi G, Floridia S, De Giorgi F, Telese R, Braccia A, Zampogna A, Pinola G, Patera M, Belluscio G, Crivellari S, Antoniazzi E, Cascino S, Giaco A, Masaracchio A, Moreschi GC, Catotti M, Eleopra R. Integrated management of atypical parkinsonism: a home-based patient-centered healthcare delivery based on telenursing-the IMPACT study protocol. Ther Adv Neurol Disord. 2025 Apr 3;18:17562864241299347. doi: 10.1177/17562864241299347. eCollection 2025. PMID 40190837